CLINICAL TRIAL: NCT01221428
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cells Infusion for Ulcerative Colitis
Brief Title: Umbilical Cord Mesenchymal Stem Cells Infusion for Ulcerative Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Wang, Yangang MD, Stem Cell Research Center of Medical School Hospital of Qingdao University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCKJ004
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-07

CONDITIONS: Ulcerative Colitis; Mesenchymal Stem Cells; Umbilical Cord
Keywords: Ulcerative colitis; Mesenchymal Stem Cells; Umbilical Cord
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord mesenchymal stem cells (Experimental): Intravenous infusion of ex vivo cultured umbilical cord mesenchymal stem cells,one week later,conduct intervention operation to inject mesenchymal stem cells to mesenteric artery.
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells — Intravenous infusion of ex vivo cultured umbilical cord mesenchymal stem cells(2*10/7),one week later,conduct intervention operation to inject mesenchymal stem cells to mesenteric artery(1*10/7).
  Other Names: Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to determine whether umbilical cord Mesenchymal Stem Cells of treatment for ulcerative colitis is safe and effective.

DETAILED DESCRIPTION:
Ulcerative colitis is characterized as chronic and nonspecific inflammation of gastroenteritis tract．Nowadays，etiology and pathogenesis of UC have been unclear．Recent basic research has been revealed that stem cell can settle down in epithelium of gastroenteritis tract，which provide a hope for treating the disease.We hope umbilical cord Mesenchymal Stem Cells could not only address the need for epithelial cell replacement but also control of the autoimmune response to mocous membrane of colon.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Ulcerative colitis described according to usual criteria.
* Refractoriness Ulcerative colitis or unefficient by using other therapy
* Signed informed consent form.

Exclusion Criteria:

* History of neoplasm or hematological disease
* Uncontrolled high blood pressure (>180/110)
* Severe cardiac insufficiency (New York Heart Association [NYHA] IV) or ejection fraction<30%
* Malignant ventricular arrythmia
* Deep venous thrombosis during the last 3 months
* Active bacterial infection
* Body mass index > 35 Kg/m2
* Stroke or myocardial infarction during the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the result of enteroscopy and pathological report | 3 months

SECONDARY OUTCOMES:
the clinical symptom (including stomachache,abdominal distention,bloody purulent stool) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Stem Cell Research Center of Medical School Hospital of Qingdao University, Qingdao, Shandong, China